CLINICAL TRIAL: NCT00407407
Title: A Phase I Dose Escalation Study of ABI-007 With Carboplatin TM as First-Line Therapy in Patients With Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Carcinoma
Brief Title: ABI-007 With Carboplatin as First-Line Therapy in Patients With Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: MTD not determined
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA034; NCT00405223 (obsolete NCT alias)
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Fallopian Tube Neoplasms; Peritoneal Neoplasms; Ovarian Neoplasms
Keywords: Epithelial ovarian; Primary peritoneal or fallopian tube carcinoma; Abraxane; Carboplatin
MeSH Terms: conditions — Fallopian Tube Neoplasms; Peritoneal Neoplasms; Ovarian Neoplasms | interventions — Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ABI-007 — 80mg/m^2 to 150mg/m^2 IV every 3 weeks
Drug: Carboplatin — 6 AUC IV every 3 weeks on the same day as ABI-007

SUMMARY:
The primary purpose of this study is to determine the maximum tolerated dose and dose-limiting toxicities (DLTs) of weekly and every 3-weeks ABI-007 in combination with carboplatin (area under the curve [AUC]=6) in patients with ovarian cancer, primary peritoneal cancer, or fallopian tube cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histological diagnosis of primary peritoneal carcinoma, fallopian tube or epithelial ovarian carcinoma (Stage III or IV) with either (optimal less than or equal to 1 cm) residual disease or suboptimal residual disease following initial appropriate surgery.
* Patients with the following histologically confirmed types of ovarian cancer are eligible: serous cystadenocarcinoma, mucinous cystadenocarcinoma, clear cell adenocarcinoma, adenocarcinoma (unspecified), malignant Brenner's tumor, endometrioid adenocarcinoma, undifferentiated carcinoma, mixed epithelial carcinoma and transitional cell carcinoma. Patients with extraovarian papillary serous cystadenocarcinoma are eligible.
* Patients who do not have measurable disease may be included and will be assessed for toxicity and progression-free survival only. Measurable disease is NOT required but when present will be followed to assess response. For patients to be evaluated for response of measurable disease, tumor must be greater than or equal to 2.0 cm with conventional computed tomography (CT) imaging or greater than or equal to 1.0 cm with spiral CT imaging.
* No prior chemotherapy for ovarian cancer is permitted.
* Patients must be entered no more than 12 weeks postoperatively.
* ECOG performance status 0-2.
* Age greater than or equal to 18 years.
* Patient has the following blood counts at Baseline:

  * ANC greater than or equal to 1.5 x 10^9 cells/L;
  * Platelets greater than or equal to 100 x 10^9 cells/L;
  * Hemoglobin (Hgb) greater than or equal to 9 g/dL.
* Patient has the following blood chemistry levels at Baseline:

  * AST (SGOT), ALT (SGPT) less than or equal to 2.5x upper limit of normal range (ULN);
  * Total bilirubin less than or equal to ULN;
  * Creatinine less than or equal to 1.5 mg/dL.
* Peripheral neuropathy Grade 0 or 1 by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE).
* It is assumed that almost all patients already had bilateral oophorectomy. However, if a female of childbearing potential, has a negative pregnancy test (within 72 hours of the first dose of study drug), the patient must agree to use an effective method to avoid pregnancy for the duration of the study.
* Patients must have signed an approved informed consent and authorization permitting the release of personal health information.

Exclusion Criteria:

* Patients who have received any prior treatment, other than initial debulking surgery, for the cancer being treated in this study. Patients may have received adjuvant chemotherapy for localized breast cancer, if the therapy was completed greater than or equal to 3 years before registration in this study and if the patient remains free of recurrent or metastatic disease.
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis. Prior radiation for localized cancer of the breast, head and neck or skin is permitted if it was completed greater than or equal to 3 years before registration in this study and if the patient remains free of recurrent metastatic disease.
* Concurrent immunotherapy or hormonal therapy for ovarian cancer.
* Parenchymal brain metastases, unless documented to be clinically and radiographically stable for at least 6 months after treatment for the disease.
* Serious intercurrent medical or psychiatric illness, including serious active infection (i.e. requiring antibiotics).
* Patients with borderline or low malignant potential tumors.
* History of other malignancy within the last 5 years, which could affect the diagnosis or assessment of ovarian cancer.
* Patients who have received an investigational drug within the previous 3 weeks.
* Patient is currently enrolled in a different clinical study in which investigational procedures are performed or investigational therapies are administered. Also, a patient may not enroll in such clinical trials while participating in this study.
* Pregnant or nursing women.
* Patients with unstable angina or those who have had myocardial infarction within the past 6 months. Patients with evidence of cardiac conduction abnormalities (e.g., bundle branch block, heart block) are eligible if their cardiac status has been stable for the 6 months prior to study entry.
* Patients with prior hypersensitivity to both Taxol and Taxotere.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-11-01 (Actual); Primary Completion 2008-02-01 (Actual); Study Completion 2008-02-01 (Actual)

PRIMARY OUTCOMES:
Primary: Safety/tolerability endpoints are the maximum tolerated dose and dose-limiting toxicities | 18 months

SECONDARY OUTCOMES:
Safety-AEs, SAEs, Lab abnormalities, incidence of patients experiencing dose modification of those interruptions &/or premature of d/c pf study drug | Patient progression or until discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Robert Coleman, MD, Principal Investigator — Univeristy of Texas, MD Anderson Cancer Center
Locations (1):
- University of Texas, MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Hafner C, Windpassinger M, Tretter EV, Rebernig KA, Reindl SM, Hochreiter B, Dekan S, Haider P, Kiss H, Klein KU, Wohlrab P. Role of mitochondrial DNA level in epidural-related maternal fever: a single-centre, observational, pilot study. BMC Pregnancy Childbirth. 2024 May 3;24(1):341. doi: 10.1186/s12884-024-06551-7. PMID 38702618